CLINICAL TRIAL: NCT01716975
Title: A Randomized, Double-blind, Placebo-controlled, Parallel, 26-Week, Phase 3 Study of 2 Doses of an Alpha-7 Nicotinic Acetylcholine Receptor Agonist (EVP-6124) or Placebo as an Adjunctive Pro-cognitive Treatment in Schizophrenia Subjects on Chronic Stable Atypical Antipsychotic Therapy
Brief Title: Study of EVP-6124 (Alpha-7 nAChR) as an Adjunctive Pro-Cognitive Treatment in Schizophrenia Subjects on Chronic Stable Atypical Antipsychotic Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: FORUM Pharmaceuticals Inc (Industry)
Collaborators: Syneos Health (Other); NeuroCog Trials, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EVP-6124-016; 2012-003209-92 (EudraCT Number)
Record Dates: First submitted 2012-10-19; First posted 2012-10-30 (Estimated); Last update posted 2016-05-03 (Estimated); Status verified 2015-06

CONDITIONS: Schizophrenia; Impaired Cognition
Keywords: Schizophrenia; Cognition; Cognition Impairment; Alpha-7 nAChR
MeSH Terms: conditions — Schizophrenia; Cognition Disorders | interventions — 7-chloro-N-quinuclidin-3-yl-benzo(b)thiophene-2-carboxamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- EVP-6124, Placebo (Placebo Comparator): Placebo, Tablet, Once Daily, Day -14 through Day 182
  Interventions: Drug: Placebo
- EVP-6124, low dose (Experimental): low dose, Tablet, Once Daily, Day 1 through Day 182
  Interventions: Drug: EVP-6124
- EVP-6124, high dose (Experimental): high dose, Tablet, Once Daily, Day 1 through Day 182
  Interventions: Drug: EVP-6124

INTERVENTIONS:
Drug: EVP-6124 — Arms 1, 2
  Arms: EVP-6124, high dose; EVP-6124, low dose
Drug: Placebo — Arm 3
  Arms: EVP-6124, Placebo

SUMMARY:
The purpose of this study is to determine if EVP-6124 (an alpha-7 nAChR agonist) enhances the cognitive abilities of subjects with Schizophrenia who are also taking stable antipsychotic therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 50 years of age, inclusive
* Signed informed consent, indicating that the subject understands the purpose of and procedures required for the study, before the initiation of any study specific procedures. Subjects who are unable to provide informed consent will not be included in the study.
* Resides in a stable living situation, according to the investigator's judgment, and must have an identified informant who should be consistent throughout the study. If possible, the informant should accompany the subject or be available for in person ratings at the screening, baseline (Day 1), and final study visits. In person informant ratings on all relevant study visits are preferred whenever possible. However, if the informant is not available for in person ratings, telephone interview is acceptable. The informant must be available for a telephone interview throughout the study at all visits. As long as both the informant visit and subject visit are within the study visit windows, it is not necessary that they occur on the same day. The informant must interact with the subject at least 2 times a week.
* Diagnosis of Schizophrenia of at least 3 years duration. This diagnosis can be established utilizing the SCID-I, direct clinical assessments, family, informants, and confirmation of diagnosis from clinical sources. These may include medical records, confirmation of diagnosis by treating clinician through telephone contact, or written confirmation from treating clinic. If the listed sources are not available, other sources of diagnostic confirmation may also be acceptable after discussion with the medical monitor.
* Treated with atypical antipsychotic drug (in any approved dosage form) other than Clozapine at a stable dose for at least 8 weeks prior to screening and be clinically stable; the subject must remain clinically stable (in the opinion of the principal investigator) through randomization. The use of up to 2 atypical antipsychotic drugs is permitted, as long as in the opinion of the investigator, the second medication is not required to control treatment-resistant or intractable psychotic symptoms. No subject will be washed off antipsychotic therapy to become eligible for this study.
* Schizophrenia clinical symptom burden severity defined by the following: a Brief Psychiatric Rating Scale (BPRS) Conceptual Disorganization item score ≤ 4; and a BPRS Hallucinatory Behavior item score ≤ 5, or an Unusual Thought Content item score ≤ 5. Either Hallucinatory Behavior or Unusual Thought Content, but not both, may have a score of 6 (but not > 6).
* Simpson-Angus Scale (SAS) total score ≤ 6
* Calgary Depression Scale for Schizophrenia (CDSS) total score ≤ 10
* General health status acceptable for participation in a 26-week clinical study
* Fertile, sexually active subjects (men and women) must use an effective method of contraception during the study
* Fluency (oral and written) in the language in which the standardized tests will be administered
* The ability to refrain from using any tobacco or other nicotine-containing products for at least 30 minutes before any cognitive testing

Exclusion Criteria:

* Hospitalization within 12 weeks before screening or during the screening period, or change of antipsychotic medication or dose within 8 weeks before screening or during the screening period.
* Participation in another therapeutic (medication administration) clinical study within the past 2 months.
* Psychiatric hospitalization or incarcerations due to breakthrough symptoms or acute exacerbations for a period of 3 months before screening. Subjects with a recent "social" hospitalization or incarceration may be entered into screening after consultation with the medical monitor
* Likelihood, in the opinion of the investigator, that either the subject or informant will be unable to complete a 26-week study
* Treatment with prohibited antipsychotic drug, and/or treatment with more than 2 permitted antipsychotic drugs. Treatment with a first-generation antipsychotic drug (typical antipsychotic) is prohibited unless it is administered at a low dose after discussion with the medical monitor
* Current treatment with any anticholinergic agent
* Diagnostic and Statistical Manual of Mental Disorders, fourth edition (DSM-IV) criteria met for alcohol abuse within the past 3 months or substance abuse (other than nicotine) within the last 6 months before screening
* Significant suicide risk as defined by 1) suicidal ideation as endorsed on items 4 or 5 of the Columbia-Suicide Severity Rating Scale (C-SSRS) within the past year; 2) suicidal behavior detected by the C-SSRS during the past 2 years, or 3) psychiatric interview and examination
* Stroke within 6 months before screening, history of brain tumor, subdural hematoma, or other clinically significant neurological condition, head trauma with loss of consciousness within 12 months before screening
* Monoamine oxidase inhibitor antidepressants or tricyclic medications used in antidepressant doses are excluded. Other antidepressant medications are allowed if the subject has been treated with a stable dose for at least 3 months before screening
* Immunosuppressants, mood stabilizers, chronic use of a sedative hypnotic drug, chronic intake of clinically significant doses of opioid containing analgesics or any current methadone treatment all in the judgment of the investigator may be permitted depending on the circumstance
* Use of Central Nervous System(CNS) stimulants
* Nicotine therapy (including patches), varenicline (Chantix), or similar therapeutic agent within the last six months before screening
* Use of a benzodiazepine medication is allowed if the subject has not had a change in medication or dose for at least 3 months. For subjects prescribed benzodiazepines, short-acting benzodiazepines are to be used whenever possible. Use of longer-acting benzodiazepines may be acceptable if prior authorization is obtained from the medical monitor. When possible, benzodiazepines should not be administered within 3 hours before cognitive testing. The use of more than one sedative-hypnotic medication is not allowed.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 767 (Actual)
Dates: Start 2012-10; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in the Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery (MCCB) to Day 182 | Baseline to Day 182 or Early Termination
Change from Baseline in the Schizophrenia Cognition Rating Scale (SCoRs) to Day 182 | Baseline to Day 182 or Early Termination
Safety and Tolerability of EVP-6124 or Placebo in Subjects with Schizophrenia | Screening (Day -42 to Day -15) to Day 182 or Early Terminiation
  All adverse experiences spontaneously reported by subject and/or observed by investigator and repeated clinical evaluation of physical examinations, vital signs, 12-lead ECG (electrocardiogram), ambulatory ECG, and laboratory tests (hematology/blood/chemistry/urinalysis)

SECONDARY OUTCOMES:
Change from Baseline in the Positive and Negative Symptom Scale (PANSS) to Day 182 | Baseline to Day 182 or Early Termination
Change from Baseline in the Clinical Global Impression-Severity (CGI-S) to Day 182 | Baseline to Day 182 or Early Termination
Change from Baseline in the Clinical Global Impression Change Scale (CGI-C) to Day 182 | Baseline to Day 182 or Early Termination
Change from Baseline in the EuroQOL-5D (EQ-5D) to Day 182 | Baseline to Day 182 or Early Termination

CONTACTS AND LOCATIONS:
Locations (106):
- United States (49):
  - Phoenixville, Arizona
  - Little Rock, Arkansas
  - Cerritos, California
  - Chino, California
  - Costa Mesa, California
  - Garden Grove, California
  - Glendale, California
  - Norwalk, California
  - Oakland, California
  - Oakland Park, California
  - Oceanside, California
  - Riverside, California
  - San Diego, California
  - San Gabriel, California
  - Santa Ana, California
  - Sherman Oaks, California
  - Washington D.C., District of Columbia
  - Bradenton, Florida
  - Miami, Florida
  - Miami Springs, Florida
  - North Miami, Florida
  - Orlando, Florida
  - Marietta, Georgia
  - Smyrna, Georgia
  - Chicago, Illinois
  - Oak Brook, Illinois
  - Oak Park, Illinois
  - Wichita, Kansas
  - Lake Charles, Louisiana
  - Shreveport, Louisiana
  - Rockville, Maryland
  - Boston, Massachusetts
  - Saint Charles, Missouri
  - St Louis, Missouri
  - Lincoln, Nebraska
  - Princeton, New Jersey
  - Jamaica, New York
  - New York, New York
  - Rochester, New York
  - Charlotte, North Carolina
  - Beachwood, Ohio
  - Oklahoma City, Oklahoma
  - Jenkintown, Pennsylvania
  - Austin, Texas
  - Dallas, Texas
  - Salt Lake City, Utah
  - Bellevue, Washington
  - Richland, Washington
  - Spokane, Washington
- Argentina (5):
  - Banfield, Buenos Aires
  - Caba, Buenos Aires F.D.
  - Mendoza, Mendoza Province
  - Rosario, Santa Fe Province
  - Santiago del Estero
- Australia (2):
  - Adelaide, South Australia
  - Mount Claremont, Western Australia
- Brazil (3):
  - Salvader, Estado de Bahia
  - Belo Horizonte, Minas Gerais
  - Curitiba, Paraná
- Colombia (4):
  - Medellín, Antioquia
  - Barranquilla, Atlántico
  - Pereira, Risaralda Department
  - Bogota D.C.
- Italy (9):
  - Florence, FL
  - Milan, MI
  - Ban
  - Barl
  - Catania
  - Lucca
  - Milan
  - Pisa
  - Roma
- Mexico (3):
  - Monterrey, Nuevo León
  - Mexico City
  - San Luis Potosí City
- Poland (8):
  - Bełchatów
  - Chełmno
  - Karakow
  - Kielce
  - Kotarbinskiego
  - Sosnowiec
  - Torun
  - Wroclaw
- Romania (7):
  - Campulung Muscel, Argeş
  - Oradea, Bihor County
  - Cluj-Napoca, Cluj
  - Palazu Mare, Constanța County
  - Iași, Iaşi
  - Târgu Mureş, Munes
  - Bucharest, Sector 4
- Russia (5):
  - Saint Petersburg, Sankt-Peterburg
  - Smolensk, Smolensk Oblast
  - Moscow
  - Samara
  - Yaroslavl
- Ukraine (7):
  - Vil. Stepanivka, Kherson Oblast
  - Dnipropetrovsk
  - Kharkiv
  - Kyiv
  - Lviv
  - Poltava
  - Vinnytsia
- United Kingdom (4):
  - Cambridge, Cambridgeshire
  - Newcastle upon Tyne, Tyne and Wear
  - Exeter
  - London